CLINICAL TRIAL: NCT00796120
Title: A Randomized, Multicenter, Phase III Trial of Trabectedin (Yondelis) Versus Doxorubicin-based Chemotherapy as First-Line Therapy in Patients With Translocation-Related Sarcomas (TRS)
Brief Title: An Efficacy and Safety Study of Trabectedin Versus Doxorubicin-Based Chemotherapy in Participants With Translocation-Related Sarcomas (TRS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015769; ET-C-002-07 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Results first posted 2014-09-16 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoma
Keywords: Sarcomas; Trabectedin; Doxorubicin; Ifosfamide; YONDELIS
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trabectedin (Experimental): Trabectedin 1.5 milligram per square meter (mg/m^2) will be given as 24-hour continuous intravenous infusion every 3 weeks until disease progression.
  Interventions: Drug: Trabectedin
- Doxorubicin plus Ifosfamide (Active Comparator): Doxorubicin (as a monotherapy) 75 mg per m^2 will be given intravenously every 3 weeks or Doxorubicin 60 mg per m^2 will be given intravenously every 3 weeks followed by ifosfamide 6 to 9 gram (g)/m^2 every 3 weeks until disease progression.
  Interventions: Drug: Doxorubicin; Drug: Ifosfamide

INTERVENTIONS:
Drug: Trabectedin — Trabectedin 1.5 milligram per square meter (mg/m^2) will be given as 24-hour continuous intravenous infusion every 3 weeks until disease progression.
  Arms: Trabectedin
Drug: Doxorubicin — Doxorubicin 60 or 75 mg/m^2 will be given intravenously every 3 weeks until disease progression.
  Arms: Doxorubicin plus Ifosfamide
Drug: Ifosfamide — Ifosfamide 6 to 9 g/m^2 will be given intravenously every 3 weeks until disease progression.
  Arms: Doxorubicin plus Ifosfamide

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of trabectedin compared to standard doxorubicin in participants with advanced translocation-related sarcomas (cancer of connective tissue cells) (TRS).

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), multicenter (when more than one hospital or medical school team work on a medical research study), Phase 3 trial to evaluate the efficacy and safety of trabectedin as compared to standard doxorubicin in participants with advanced TRS. Participants will be randomized in a 1:1 ratio to either of the 2 treatment groups, that is, trabectedin or doxorubicin plus ifosfamide group. Participants in trabectedin group will receive trabectedin 1.5 milligram per square meter (mg/m^2) given as a 24-hour continuous intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) every 3 weeks and in doxorubicin plus ifosfamide group participants will receive doxorubicin 60 or 75 mg/m^2 intravenously every 3 weeks followed by ifosfamide 6 to 9 gram (g)/m^2 every 3 weeks. Participants in either treatment arm will continue receiving therapy in the absence of progressive disease (PD) or intolerable side effects, until the participants' consent is withdrawn or the eligibility criteria for continuing treatment are no longer fulfilled, or when a concurrent condition precludes continuation of treatment. Efficacy will be assessed primarily by evaluating progression-free survival (PFS). Participants' safety will be monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of translocation-related sarcomas (TRS) including the following subtypes: alveolar soft part sarcoma, angiomatoid fibrous histiocytoma, clear cell sarcoma, desmoplastic small round cell tumor, low grade endometrial stromal sarcoma (prior hormone therapy allowed), low grade fibromyxoid sarcoma, myxoid chondrosarcoma, myxoid/round cell liposarcoma (MRCL) and synovial sarcoma
* Participants must have unresectable locally advanced or metastatic progressive disease prior to enrolment
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2
* Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) within normal limits according to institutional standards, as shown by echocardiography or scintigraphy multiple-gated acquisition scan [MUGA]
* Measurable disease as defined by the radiological (computed tomography [CT] scan and magnetic resonance imaging [MRI]) Response Evaluation Criteria in Solid Tumors (RECIST v.1.0) guidelines

Exclusion Criteria:

* Known hypersensitivity to any components of the intravenous formulation of trabectedin or the comparators
* Prior chemotherapy treatment or irradiation of the lesion if only one target lesion is available
* Brain metastases and/or leptomeningeal metastases, even if treated
* Pregnant or lactating women or men and women of reproductive potential who are not using effective contraceptive methods
* History of another neoplastic disease (except basal cell carcinoma or cervical carcinoma in situ adequately treated) unless in remission for five years or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, LLC Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (21):
- United States (6):
  - Santa Monica, California
  - Boston, Massachusetts
  - Albuquerque, New Mexico
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Salt Lake City, Utah
- France (5):
  - Boreaux
  - Lille
  - Lyon
  - Paris
  - Villejuif
- Germany (3):
  - Bad Saarow
  - Cologne
  - Mannheim
- Spain (3):
  - Barcelona
  - Palma
  - Valencia
- United Kingdom (4):
  - Edinburgh
  - Glasgow
  - London
  - Manchester

REFERENCES:
- [Derived] Blay JY, Leahy MG, Nguyen BB, Patel SR, Hohenberger P, Santoro A, Staddon AP, Penel N, Piperno-Neumann S, Hendifar A, Lardelli P, Nieto A, Alfaro V, Chawla SP. Randomised phase III trial of trabectedin versus doxorubicin-based chemotherapy as first-line therapy in translocation-related sarcomas. Eur J Cancer. 2014 Apr;50(6):1137-47. doi: 10.1016/j.ejca.2014.01.012. Epub 2014 Feb 7. PMID 24512981

RESULTS

PARTICIPANT FLOW:
Groups:
- Trabectedin: Trabectedin 1.5 milligram per square meter (mg/m^2) given as 24-hour continuous intravenous infusion every 3 weeks until disease progression.
- Doxorubicin Plus Ifosfamide: Doxorubicin (as a monotherapy) 75 mg per m^2 will be given intravenously every 3 weeks or Doxorubicin 60 mg per m^2 will be given intravenously every 3 weeks along with ifosfamide 6 to 9 gram (g)/m^2 every 3 weeks until disease progression.
Period: Overall Study
Arm/Group | Trabectedin | Doxorubicin Plus Ifosfamide
Started | 61 | 60
Treated | 61 | 57
Completed | 0 | 0
Not Completed | 61 | 60
Not completed — Death | 3 | 0
Not completed — Adverse Event | 11 | 6
Not completed — Progressive disease | 22 | 13
Not completed — Participant refusal | 3 | 4
Not completed — Other | 6 | 17
Not completed — Physician Decision | 16 | 17
Not completed — Randomized but not treated | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trabectedin | Doxorubicin Plus Ifosfamide | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Customized [Number; unit: participants]
  >=18 to <=49 years | 33 | 30 | 63
  >=50 to <=65 years | 19 | 21 | 40
  >=65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Progression - Free Survival (PFS)
Description: The PFS was assessed as median number of days from the date of randomization until the first documented sign of disease progression (increase in disease; radiographic, clinical, or both) or death due to any cause, whichever occurred earlier.
Time Frame: Every 6 weeks from randomization during the first 9 months and thereafter, every 9 weeks up to 20 months
Population: Efficacy population included all participants randomly assigned to either treatment arm with externally confirmed pathological and molecular diagnosis of translocation-related sarcomas (TRS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trabectedin | Doxorubicin Plus Ifosfamide
Number analyzed (Participants) | 51 | 37
months | 19.6 [5.7 to 32.3] | 8.3 [7.1 to 25.0]

2. Secondary Outcome: 6-month Progression - Free Survival
Description: Percentage of participants survived for 6 months from the start of study treatment without progression of disease. Progression of the disease was associated with increasing symptoms, including pain from new or progressing lesions. Delay in disease progression generally represents a clinical benefit to the participant.
Time Frame: 6 months
Population: Efficacy population included all participants randomly assigned to either treatment arm with externally confirmed pathological and molecular diagnosis of TRS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trabectedin | Doxorubicin Plus Ifosfamide
Number analyzed (Participants) | 51 | 37
percentage of participants | 66.7 [50.6 to 82.8] | 78.3 [64.0 to 92.5]

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Tumor response was assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Partial Response (PR)=at least 30% reduction in the sum of the longest dimensions (LD) of all target lesions in reference to the baseline sum LD, Complete Response (CR) =Disappearance of all non-target lesions. Percentage of participants with objective tumor response was determined by the number of participants with PR or CR divided by the total number of response-evaluable participants.
Time Frame: Every 6 weeks during first 9 months of the study and thereafter every 9 weeks up to 20 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trabectedin | Doxorubicin Plus Ifosfamide
Number analyzed (Participants) | 51 | 37
percentage of participants | 5.9 [1.2 to 16.2] | 27.0 [13.8 to 44.1]

4. Secondary Outcome: Overall Survival
Description: Overall survival defined as time from the date of randomization to the date of death. For participants who were alive at the time of analysis, overall survival was censored at the last contact date.
Time Frame: Baseline up to End of Study (an average of 4 years)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trabectedin | Doxorubicin Plus Ifosfamide
Number analyzed (Participants) | 51 | 37
months | 46.6 [27.5 to NA] — Upper limit of confidence interval was not reached because of high censorship rate that is smaller number of events. | 33.5 [21.6 to NA] — Upper limit of confidence interval was not reached because of high censorship rate that is smaller number of events.

5. Secondary Outcome: Duration of Response (DOR)
Description: The DOR is defined as the time from date of first documentation of response (CR or PR, whichever comes first) to the date of documented PD or death. PR=at least 30% reduction in the sum of the longest dimensions (LD) of all target lesions in reference to the baseline sum LD, CR =Disappearance of all non-target lesions.
Time Frame: Up to 20 months
Population: Efficacy population included all participants randomly assigned to either treatment arm with externally confirmed pathological and molecular diagnosis of TRS. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Trabectedin | Doxorubicin Plus Ifosfamide
Number analyzed (Participants) | 3 | 10
days | NA [7.0 to NA] — Median and upper confidence interval point estimates were not reached because of high censorship rate that is smaller number of events. | NA [4.4 to NA] — Median and upper confidence interval point estimates were not reached because of high censorship rate that is smaller number of events.

ADVERSE EVENTS:
Arm/Group | Trabectedin | Doxorubicin Plus Ifosfamide
Serious Adverse Events (participants affected / at risk) | 24/61 | 16/57
Other Adverse Events (participants affected / at risk) | 55/61 | 52/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=61) | Doxorubicin Plus Ifosfamide (N=57)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Hypothermia (General disorders) | 1 | 0
Injection site extravasation (General disorders) | 3 | 0
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 2
Liver injury (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 4 | 0
Device related infection (Infections and infestations) | 3 | 0
Erysipelas (Infections and infestations) | 1 | 0
Infusion site infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumococcal bacteremia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Blood CPK increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dyspraxia (Nervous system disorders) | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=61) | Doxorubicin Plus Ifosfamide (N=57)
Anaemia (Blood and lymphatic system disorders) | 11 | 13
Neutropenia (Blood and lymphatic system disorders) | 29 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 2
Tachycardia (Cardiac disorders) | 3 | 4
Eye irritation (Eye disorders) | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 8 | 5
Constipation (Gastrointestinal disorders) | 27 | 16
Diarrhoea (Gastrointestinal disorders) | 15 | 15
Dry mouth (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 8 | 7
Haemorrhoids (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 46 | 40
Oral pain (Gastrointestinal disorders) | 0 | 10
Stomatitis (Gastrointestinal disorders) | 1 | 6
Vomiting (Gastrointestinal disorders) | 29 | 16
Chest pain (General disorders) | 3 | 3
Fatigue (General disorders) | 45 | 42
Mass (General disorders) | 10 | 5
Mucosal inflammation (General disorders) | 4 | 15
Oedema peripheral (General disorders) | 18 | 6
Pain (General disorders) | 2 | 3
Pyrexia (General disorders) | 10 | 11
Candidiasis (Infections and infestations) | 0 | 3
Catheter related infection (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Alanine aminotransferase increased (Investigations) | 19 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 0
Blood alkaline phosphataseincreased (Investigations) | 6 | 0
Blood creatine phosphokinase increased (Investigations) | 4 | 1
Gamma-glutamyltransferase increased (Investigations) | 6 | 0
Weight decreased (Investigations) | 4 | 8
Anorexia (Metabolism and nutrition disorders) | 20 | 15
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 9
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 | 33
Dizziness (Nervous system disorders) | 5 | 7
Dysgeusia (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 13 | 14
Neuropathy peripheral (Nervous system disorders) | 4 | 0
Paraesthesia (Nervous system disorders) | 2 | 3
Tremor (Nervous system disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 12 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 25
Rash (Skin and subcutaneous tissue disorders) | 4 | 6
Scar (Skin and subcutaneous tissue disorders) | 4 | 2
Deep vein thrombosis (Vascular disorders) | 4 | 0
Hypertension (Vascular disorders) | 7 | 0
Hypotension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before Investigators of this study publicly disclose information, PharmaMar must be provided with at least 60 days to review and approve disclosure in order to ensure that confidential and proprietary data are protected. If PharmaMar determines that patentable patient matter is disclosed in the proposed disclosure, the latter shall be withheld for period of time considered convenient.